CLINICAL TRIAL: NCT05142163
Title: Stroke Volume Variation and Plethysmography Variability Index as Goal Directed Fluid Therapy in Major Oncosurgeries
Acronym: SVV PVI GDFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Dr Anita Kulkarni, Senior Consultant, Rajiv Gandhi Cancer Institute & Research Center, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RGCI/GDFT
Record Dates: First submitted 2021-11-06; First posted 2021-12-02 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Goal Directed Fluid Therapy
Keywords: Goal directed Fluid Therapy; Stroke Volume Variation; Plethysmography

STUDY DESIGN:
Intervention Model Description: Patients were allotted to either SVV Guided or PVI Guided Intraoperative Fluid Therapy
Who Masked: Participant
Masking Description: Patient were masked about belonging to SVV Guided or PVI Guided Group to receive Intraoperative Fluid Therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroke Volume Variation Guided Fluid Therapy (Active Comparator): Patients will receive maintenance Fluids as crystalloids intraoperative to maintain SVV <11%, for values >11%colloid bolus 6%hydroxyethyl starch will be given and fluid responsiveness noted.
  Interventions: Other: Intraoperative SVV Guided Fluid Therapy
- Plethysmography Variability Index Guided Fluid Therapy (Active Comparator): Patients will receive maintenance Fluids as crystalloids intraoperative to maintain PVI <11%, for values >11%colloid bolus 6%hydroxyethyl starch will be given and fluid responsiveness noted.
  Interventions: Other: Intraoperative PVI Guided Fluid Therapy

INTERVENTIONS:
Other: Intraoperative SVV Guided Fluid Therapy — Patients will receive intraoperative maintenance Fluids as crystalloids to maintain SVV <11%, for values >11%colloid bolus 6%hydroxyethyl starch will be given and fluid responsiveness noted.
  Arms: Stroke Volume Variation Guided Fluid Therapy
Other: Intraoperative PVI Guided Fluid Therapy — Patients will receive intraoperative maintenance Fluids as crystalloids to maintain PVI <10%, for values >10%colloid bolus 6%hydroxyethyl starch will be given and fluid responsiveness noted.
  Arms: Plethysmography Variability Index Guided Fluid Therapy

SUMMARY:
Patients were allotted to two Groups , SVV Guided Fluid Therapy Group received intraoperative fluids to maintain SVV <11 , and PVI Guided Group received intraoperative Fluids to maintain PVI<11

DETAILED DESCRIPTION:
Preinduction Epidural catheter will be placed and Standard General Anaesthesia with Volume Controlled Ventilation (Tidal Volume 8ml/Kilogram ) and Positive End Expiratory Pressure 5 centimeters of water for all patients. Postinduction Radial artery cannulation and Ultrasound guided Internal Jugular cannulation will be performed for all patients .Maintenance Fluid crystalloids 2ml/kg will be given to both the Groups. In Stroke Volume Variation SVV Group Flotrac Transducer (MHD8 model Edwards Lifesciences LLC, Irvine,CA 92614,USA) will be attached to radial artery cannula to obtain SVV values and for values > 11 colloid bolus 200ml will be given over 10 minutes and postbolus values noted. In Plethysmography Variability Index PVI Group pulse Oximeter will be placed on index finger and covered to avoid ambient light will be attached to Masimo Radical 97 Monitor to measure continuous Perfusion Index and Plethysmography Variability Index for values >11 colloid bolus 200ml will be given over 10 minutes and change in PVI value noted. Intraoperative heart rate , Mean arterial Pressure , Oxygen Saturation, End tidal carbon dioxide, Central venous pressure , Urine output will be measured in all patients.With optimal fluids if Mean Arterial Pressure is below 70 mmHg than titrating dosage Norepinephrine infusion will be commenced.At the end of surgery reversal agents will be administered and trachea extubated , note will be made of any patient requiring postoperative ventilator support.Arterial blood gas analysis will be performed at beginning and end of surgery and at postoperative 24 and 48 hours to measure serum lactate levels . Patient will be monitored in Postanaesthesia Care Unit for any Cardiac , Respiratory event , Serum Creatinine levels will be measures at 24 and 48 hours , Appearance of bowel sounds will be noted , Length of ICU stay will be recorded for all patients.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing Open major Oncosurgeries under General Anaesthesia

Exclusion Criteria

Patient Refusal

Left ventricular Ejection Fraction <40%

Cardiac arrythmias

Severe valvular heart disease

Peripheral Vascular Disease

Laparoscopic surgeries

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
To compare Total intraoperative Fluid requirement in millilitres and Fluid Responsiveness in SVV and PVI Group. | upto 8 hours
  Patients in SVV Group will receive Crystalloids and colloid bolus 200ml to maintain SVV <11 .Patients in PVI Group will receive Crystalloids and colloid bolus to maintain PVI<11, Postbolus response to SVV and PVI values will be noted.

SECONDARY OUTCOMES:
To Measure Serum Lactate levels mmol/L in SVV and PVI Group. | upto 72 hours postoperative
  Intraoperative at beginning and end of surgery and upto 72 hours serum Lactate levels will
  be measured.
Postoperative Cardiac complication | upto72 hours
  Requirement of Inotrope Nonadrenaline
Postoperative Respiratory complication | upto 72 hours
  Ventilator support
Postoperative Renal complication | upto72 hours
  Increase serum creatinine values
Length of ICU stay | upto72 hours
  Duration in hours stay in PACU

CONTACTS AND LOCATIONS:
Overall Officials: Anita Kulkarni, MD, Principal Investigator — Senior Consultant
Locations (1):
- Rajiv Gandhi Cancer Institute and Research Centre, Delhi, India

IPD SHARING:
Plan to Share IPD: No